CLINICAL TRIAL: NCT02850224
Title: Pediatric Preventative Health Screenings - Obesity and Family-Centered
Brief Title: Pediatric Preventative Health Screenings - Obesity and Family-Centered Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Andrea Cassidy-Bushrow, PhD, Associate Scientist, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: B21201
Record Dates: First submitted 2016-06-30; First posted 2016-07-29 (Estimated); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Obesity; Overweight; Blood Pressure; Hypercholesteremia; Diabetes
MeSH Terms: conditions — Obesity; Overweight; Hypercholesterolemia; Diabetes Mellitus | interventions — Motivational Interviewing; Patient Outcome Assessment

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational interviewing to elicit PCO in pediatrics (Experimental): Providers will be randomized into a patient-centered outcomes (PCO) education course or standard of care. The PCO education course will educate and test providers on patient-centered outcomes of interest and appropriate methods to deliver PCO care.
  Providers randomized into the intervention arm will be required to take a brief, one-hour, webinar describing the background, problem, results from focus groups we conducted, and a training program on motivational interviewing. After completing the course, providers will be required to complete an evaluation.
  Interventions: Behavioral: Motivational interviewing to elicit PCO in pediatrics
- No Intervention (No Intervention): Standard care

INTERVENTIONS:
Behavioral: Motivational interviewing to elicit PCO in pediatrics — A motivational interviewing style webinar. Physicians watch the webinar, incorporate communication techniques.
  Other Names: Motivational Interviewing; Patient-Centered Outcomes
  Arms: Motivational interviewing to elicit PCO in pediatrics

SUMMARY:
In 2012, an Expert Panel of the National Heart Lung and Blood Institute published guidelines on cardiovascular health and risk reduction in children; among these guidelines were screening recommendations for obesity and obesity-related conditions. Following publication of this report there was a call for caution and for increased patient (parent, child) input on implementing these guidelines. There are limited current studies evaluating patient-centered outcomes (PCO) in the well-child setting, however, given the childhood obesity epidemic, there is a clear need for such an evaluation. The city of Detroit, MI ranks first among 22 cities with data for the prevalence of overweight and obese youth (39.7%), making Henry Ford Health System, which is located in Detroit, MI, an ideal setting to study childhood obesity related research questions.

DETAILED DESCRIPTION:
Within this patient population, our specific aims therefore are to (1) examine current trends in screening and management of obesity and obesity-related conditions in a real-world urban practice setting; (2) examine the family (patient and parent/guardian) and clinician preferences for the identification and management of obesity and obesity-related conditions; and (3) design and conduct a Phase II pragmatic cluster randomized trial (PCRT) of an educational intervention in providers for guiding screening for obesity and obesity-related conditions during the well-child visit that incorporates and leverages PCO. Staff dedicated solely to this project will partner with the Henry Ford Health System's proposed Patient-Centered Outcomes Research Center's Cores staff members to design, execute and disseminate study results in order to affect clinical care. By seeking to understand the current screening patterns in pediatrics and by creating an education intervention for providers aimed at taking a patient/family centered approach to these preventative health screenings, we may increase PCOs which in turn may have meaningful implications for future adult health.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 2 and 18
* Henry Ford Health System Patient
* Well-child visit with participating provider
* Fluent in English

Exclusion Criteria:

* Unable to provide consent

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 703 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2018-02-19 (Actual); Study Completion 2020-07-27 (Actual)

PRIMARY OUTCOMES:
Number of participants with improved patient-centered outcomes (physical, social, and emotional health) as assessed by the PROMIS 25. | 6 weeks
Number of participants with improved health-related quality of life as assessed by the PEDsQL. | 6 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Andrea E Cassidy-Bushrow, PhD, Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No